CLINICAL TRIAL: NCT00977483
Title: Assessment of Efficacy and Safety of Thioctic Acid in the Oral Treatment of Diabetic Polyneuropathy (Stage 1 or 2) NATHAN1 A Randomized, Placebo-controlled, Double-blind Multi-centre Trial With 2 Parallel Groups
Brief Title: Assessment of Efficacy and Safety of Thioctic Acid in the Oral Treatment of Diabetic Polyneuropathy (Stage 1 or 2)
Acronym: NATHAN1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: Clinquest, Inc. (Industry); Ergomed (Industry); Quintiles, Inc. (Industry)
Responsible Party: Dr. Joachim Maus, MEDA Pharma GmbH & Co. KG
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-20557-3011; NATHAN1; D-20557/9353000001
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2016-11

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: Thioctic Acid (Experimental): 600mg tablet Thioctic Acid (alpha-lipoic acid) once daily throughout the trial
  Interventions: Drug: Thioctic Acid
- Drug: Placebo (Placebo Comparator): 1 tablet once daily throughout the trial
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thioctic Acid — 600mg tablet once daily 4 years double-blind treatment period
  Other Names: alpha-lipocic acid
  Arms: Drug: Thioctic Acid
Drug: Placebo — 1 tablet once daily 4 years double-blind treatment period
  Arms: Drug: Placebo

SUMMARY:
To assess clinical efficacy and safety of long-term orally administered thioctic acid in the treatment of diabetic polyneuropathy.

DETAILED DESCRIPTION:
Stage 1 or 2a diabetic (poly)neuropathy (DNP) (Appendix 3) in patients with diabetes mellitus (type I or II); neuropathy impairment score of the lower limbs, enlarged by 7 objective items (NISLL+7) ≥ 97.5 percentile (corresponding to 4.43 score points); total symptoms score of the feet (TSSfeet) ≤ 5.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent. Patients must have willingness and complete competence to cooperate and language barriers must not preclude adequate understanding
2. Diabetes mellitus (Type I or II), as defined by the American Diabetes Association 1997, lasting > 1 year
3. Males or females 18 to 64 years (older patients are excluded because of age-related changes in reflexes, quantitative sensory testing endpoints, and nerve conduction endpoints)
4. Patient must have a symmetric sensory-motor peripheral polyneuropathy attributable to diabetes mellitus following a thorough evaluation for other causes of neuropathy determined by performing complete medical and neurological examinations including physical and neurological history, history of medications, history of exposure to other toxins, and laboratory studies
5. Severity of diabetic polyneuropathy must be Stage 1 or 2a
6. Insulin regimen, weight, diet, and activity level must be relatively stable in the opinion of the investigator (for example, HbA1C must not vary by more than ± 2 Vol.% within 6 months preceding the study i.e. if the index measure = 10% the range would be 8-12%)
7. NIS[LL]+7 tests ≥ 97.5 percentiles (corresponding to 4.43 transformed score points)
8. NIS[LL] ≥ 2 points (NIS[LL] is based on questions 17-24, 28, 29, 34, 35, and 37 of the NIS)
9. One of the following:

   * an abnormality of nerve conduction attributes in two separate nerves, i.e. ≥99th percentile for DL or ≤1st percentile for NCV or amplitude or
   * an abnormality of HRDB, i.e. ≤ 1st percentile
10. TSS (feet) ≤5
11. Females must either be surgically sterilised (tubal ligation, bilateral oophorectomy, or hysterectomy) or at least 1 year postmenopausal or practicing an acceptable method of contraception, including oral contraceptives with a stable regimen for at least two months, depo-medroxyprogesterone, a barrier method alone (diaphragm, condoms, or contraceptive sponge with spermicidals), or an IUD that has been in place for at least two months

Exclusion Criteria:

1. Patients with proximal asymmetric neuropathy, cranial neuropathies, truncal radiculopathy, pan dysautonomia, diabetic plexopathies, or acute or active mononeuropathies (including cranial neuropathies, post-herpetic neuralgias, etc.), the presence of which might obscure accurate assessment of severity of the diabetic polyneuropathy under assessment, with the exception of carpal tunnel syndrome (CTS) or tardy ulnar neuropathy (TUN) or both
2. Neuropathy of any cause other than diabetes mellitus which might interfere with the assessment of the severity of dPNP Other neurologic diseases that may produce weakness, sensory loss, or autonomic symptoms or test abnormality which might interfere with the assessment of the severity of dPNP Myopathy of any cause which might interfere with the assessment of the severity of dPNP
3. Peripheral vascular disease severe enough to cause intermittent claudication or ischemic ulcers or limb ischemia
4. Patients with a history of ophthalmological findings suggesting a high risk for visual loss i.e., significant maculopathy or proliferative retinopathy
5. Psychiatric, psychological, or behavioural symptoms that would interfere with the patient's ability to participate in the trial
6. Patients with any active neoplastic disease except basal cell carcinoma
7. Patients with atrial fibrillation unless controlled and stabilised by medication (changed to this criterion by Amendment 1)
8. Patients with clinically significant cardiac, pulmonary, gastrointestinal, hematologic, or endocrine disease (other than diabetes) that may confound interpretation of the study results or prevent the patient from completing the study
9. Patients who have had organ transplants of any kind
10. Patients with significant hepatic or renal disease (ASAT or ALAT >2 times normal, serum creatinine >1.8 mg/dL (>159 µmol/l) for males or >1.6 mg/dL (>141 µmol/l) for females)
11. Patients with a recent history (within last 12 months) of drug or alcohol abuse
12. Use of any investigational drug within the last 6 months
13. History of severe or anaphylactic reaction to multiple drugs, sulfur products, or biologic products (changed to this criterion by Amendment 1)
14. Ketoacidosis or hypoglycaemia within last 3 months resulting in hospital admission
15. Antioxidant therapy (vitamins E > 400IU, C > 200mg, and beta-Carotene > 30mg) or pentoxyphylline within last 1 month before start of trial
16. Use of evening primrose oil or any other gamma-linolenic acid containing substance within the last 3 months
17. Use of thioctic acid > 50mg/day within last 3 months
18. History of use of medications or vitamins known to cause peripheral neuropathy including but not limited to use of phenytoin or carbamazepine over 15 or more years, or use of pyridoxine > 100mg/d within the past 12 months
19. Bilateral sural nerve biopsies
20. Existing foot ulcers
21. Pregnant or lactating females
22. Continued use of medications listed in protocol 6.3.3 (first paragraph)
23. Medication non-compliance (deviation of more than ±10% of dosages to be taken (1 tablet/day))

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 460 (Actual)
Dates: Start 1998-05; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Primary efficacy variable: Absolute change in the neuropathy impairment score lower limbs enlarged by 7 objective items (NISLL+7) between baseline (mean of Visit 0.3 and 0.4 or last available value before randomisation, respectively) and endpoint | 4 years

SECONDARY OUTCOMES:
NIS, NSC, TSS, LLF, QST, VDT, CDT and HP, QAE by means of the HRDB, amplitude CMAP, DL and MNCV on peroneal and tibial nerves, amplitude SNAP and latency on sural nerve, foot inspection, efficacy. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter James Dyck, Principal Investigator — Mayo Clinic, Dept. of Neurology, 200 First Street Southwest, Rochester, MN 55905, USA
Locations (38):
- United States (25):
  - ´Diabetes Care Center, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Medical Building, Long Beach, California
  - UCSD Neuromuscular Research Program, San Diego, California
  - University of California, San Francisco, California
  - Diabetes Research Center, Tustin, California
  - Loyola University Medical Center, Maywood, Illinois
  - Beth Israel Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Health Partners Riverside Neurology Clinic, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Missouri Dept. of Neurology, Columbia, Missouri
  - Creighton University Diabetes Center, Omaha, Nebraska
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Ney York Hospital Cornell Med Center, New York, New York
  - East Carolina University, School of Medicine, Greenville, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - University of Texas South Western Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Diabetes & Glandular Disease Center, San Antonio, Texas
  - Leonard R. Strelitz Diabetes Institutes, Norfolk, Virginia
- Croatia (2):
  - University Clinic for Diabetes, Endocrinology and Metabolic, Zagreb
  - University Clinic of Internal Medicine, Zagreb
- University Hospital, Hvidovre, Denmark
- Hospital Jean Verdler, Bondy, France
- Italy (3):
  - Policlinic University, Napoli
  - Hospital Geriatrico Diabetological Service, Padua
  - Hosptal of Parma Department of Medicine, Parma
- University Hospital Utrecht Department of Internal Medicine, Utrecht, Netherlands
- Spain (3):
  - Hospital del Mar Department Neurophysiology, Barcelona
  - Hospital Clinico y Provincial, Barcelona
  - C.H.U.S. General Hospital, Santiago de Compostela
- University Clinic, Malmo, Sweden
- Manchester Royal Infirmary Department of Medicine, Manchester, United Kingdom

REFERENCES:
- [Derived] Ziegler D, Low PA, Litchy WJ, Boulton AJ, Vinik AI, Freeman R, Samigullin R, Tritschler H, Munzel U, Maus J, Schutte K, Dyck PJ. Efficacy and safety of antioxidant treatment with alpha-lipoic acid over 4 years in diabetic polyneuropathy: the NATHAN 1 trial. Diabetes Care. 2011 Sep;34(9):2054-60. doi: 10.2337/dc11-0503. Epub 2011 Jul 20. PMID 21775755